CLINICAL TRIAL: NCT03940833
Title: Clinical Research of Adoptive BCMA CAR-NK Cells on Relapse/Refractory MM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asclepius Technology Company Group (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AsclepiusTCG02
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-tumor response of BCMA CAR-NK-92 (Experimental): Patients with relapsed and refractory MM of BCMA expression will be treated with BCMA CAR-NK 92 cells.
  Interventions: Biological: BCMA CAR-NK 92 cells

INTERVENTIONS:
Biological: BCMA CAR-NK 92 cells — The subject will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
The purpose of this study is to infuse BCMA CAR-NK 92 cells to the patients with relapsed and refractory multiple myeloma (MM), to assess the safety and feasibility of this strategy. The CAR enables the NK-92 cells to recognize and kill the MM cells by targeting of BCMA, a protein expressed of the surface of the malignant plasma cells in MM patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 80 years, expected survival > 3 months
2. Confirmed diagnosis of active MM as defined by IMWG. BCMA expression of the malignant cells must be detected by immunohistochemistry or by flow cytometry
3. BCMA-expressing B cell malignancy must be assured and must be relapsed or refractory disease
4. ECOG performance status of 0 - 1
5. Cardiac function: 1 - 2 levels; Liver: TBIL ≤ 3ULN，AST ≤ 2.5 ULN，ALT ≤ 2.5ULN; kidney: Cr ≤ 1.25ULN
6. No serious allergic constitution
7. No other serous diseases that conflicts with the clinical program
8. No other cancer history
9. Female participants of reproductive potential must have a negative serum pregnancy test
10. Subjects must have signed written, informed consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive
3. Active hepatitis B or hepatitis C infection
4. Recent or current use of glucocorticoid or other immunosuppressor
5. Serious mental disorder
6. With severe cardiac, liver, renal insufficiency, diabetes and other diseases
7. Participate in other clinical research in the past three months
8. Previously treatment with any gene therapy products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.03 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Wuxi People's Hospital, Nanjing Medical University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng YY, Du Z, Zhang X, Chng WJ, Wang S. CXCR4 and anti-BCMA CAR co-modified natural killer cells suppress multiple myeloma progression in a xenograft mouse model. Cancer Gene Ther. 2022 May;29(5):475-483. doi: 10.1038/s41417-021-00365-x. Epub 2021 Sep 1. PMID 34471234